CLINICAL TRIAL: NCT06166199
Title: Effects of High-intensity Interval Training Combined With Resistance Training in Patients With Systemic Lupus Erythematosus
Brief Title: Effects of High-intensity Interval Training in Patients With Systemic Lupus Erythematosus
Acronym: SLE-HIIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Swedish Rheumatism Association (Unknown); Region Örebro County (Other); County Council of Norrbotten, Sweden (Other Government); Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Carina Boström, Associate professor, university lecturer, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-05523-01
Record Dates: First submitted 2023-11-22; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Physical exercise; High-intensity interval training; Resistance training; Quality of life; Aerobic capacity; Fatigue; Disease activity; Patients experiences; Inflammatory markers; Muscle function; Depressive symptoms
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Motor Activity; Fatigue; Depression | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: This is a randomised-controlled single blinded multicenter study. The trial will follow the Consolidated Standards of Reporting Trials, www.consort-statement.org and comprise two arms.
  After information of the study and written informed consent, the patients are block-randomised (from the aerobic capacity results) to either an intervention group doing supervised high-intensity interval training combined with resistance training or a control group. Both groups receive standard care.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessors are blinded for which patient is randomised to which group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity interval training (HIIT) combined with resistance training (Experimental): Patients with SLE will undergo supervised HIIT on an ergometercycle 4 x 4 minutes interval (85-90% of maximal heart rate in 4 minutes and lower intensity for another 4 minutes etc). The HIIT is combined with resistance exercises for upper and lower extremity. In total the supervised training takes around 50 minutes per occasion and will be performed 2 times/week, for 3 months. In addition, the patients will exercise, according to the program, by themselves once a week.
  Between months 3 and 6 the patients exercise by themselves, 3 times/week, with video-call/telephone support from a physiotherapist once a week.
  Interventions: Behavioral: HIIT combined with resistance training
- Control group (No Intervention): Both the control group and the HIIT combined with resistance training group receive standard care.

INTERVENTIONS:
Behavioral: HIIT combined with resistance training — Patients with SLE will undergo supervised HIIT on an ergometercycle, 4 x 4 minutes interval, (85-90% of maximal heart rate in 4 minutes and lower intensity for another 4 minutes etc). The HIIT is combined with resistance exercises for upper and lower extremity. In total the training takes around 50 minutes per occasion and will be performed 2 times/week, for 3 months. In addition, the patients will exercise, according to the program, by themselves once a week.
  Between months 3 and 6 the patients exercise by themselves, 3 times/week, with video-call/telephone support from a physiotherapist once a week.
  Arms: High-intensity interval training (HIIT) combined with resistance training

SUMMARY:
The aim of this study is to evaluate the safety and effects of high-intensity interval training (HIIT) combined with resistance training in patients with systemic lupus erythematosus

DETAILED DESCRIPTION:
The overall aim of this randomized controlled study, is to evaluate the safety and effects of HIIT combined with resistance exercises on aerobic capacity, muscle function, patient reported outcomes, disease activity and immune function in patients with SLE with low to moderate disease activity and no to little organ damage. The aim is also to explore and describe patient's experiences of the training.

The research questions are:

1. What are the differences between the HIIT combined with resistance exercises and a control group, after 3 months of supervised training and after further 3 months of self training with video-call/telephone support until 6 months follow up, regarding aerobic capacity, muscle function, physician and patient reported disease activity, fatigue, depressive symptoms, and quality of life?
2. What are the differences between the HIIT combined with resistance exercises and a control group, after 3 months of supervised training and after further 3 months of self training with video-call/telephone support until 6 months follow up, regarding inflammatory markers such as interleukin 6 and 10 and interferon molecules? Both acute exercise test (maximal ergometercycle test) effects as well as the long term effects of training will be evaluated.
3. How do individuals with SLE experience HIIT combined with resistance exercises ? What are the perceived barriers and facilitators for performing and maintaining such training?

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Fulfilment of the 1982 American College of Rheumatology (ACR) criteria; or 2012 Systemic Lupus International Collaborating Clinics (SLICC/ACR-Damage Index (DI)) classification criteria; or EULAR/ACR criteria; or patients that have received the diagnosis SLE on clinical grounds
* Low to moderate disease activity, for example defined as a score of ≤5 in the clinical version of the SLE Disease Activity Index 2000 (SLEDAI-2K), i.e., excluding the serological descriptors (anti-dsDNA positivity and low complement levels)
* Low/minimal or no organ damage, for example defined as a score of ≤3 in the SLICC/ACR DI
* Stable pharmacological treatment
* The ability to perform a maximal ergometercycle exercise test
* Be able to read and understand Swedish

Exclusion Criteria:

* Symptoms or signs of cerebro-vascular disease, pulmonary embolus, pulmonary hypertension, pulmonary fibrosis, cardiovascular disease, angina pectoris, myocardial infarction, dyspnea at rest, uncontrolled blood pressure and uncontrolled diabetes within one year prior to study entry. Chronic kidney disease with
* Patients who fulfil the absolute contraindications for maximal exercise testing according to American Heart Association
* Patients who cannot perform a maximal ergometercycle exercise test due to the disease
* Diseases or other conditions that strongly reduce the ability to exercise or that exercise is not recommended
* Patients who perform regular aerobic fitness training and muscle strength exercise sessions at fixed times, >1 time/week
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Aerobic capacity | Baseline, months 3 and 6
  Aerobic capacity is measured as maximal oxygen uptake when performing a maximal symptom-limited, ergometercycle exercise test
Physical capacity | Baseline, months 3 and 6
  Physical capacity are measured when performing a symptom-limited, ergometercycle exercise test

SECONDARY OUTCOMES:
Muscle function upper extremity | Baseline, months 3 and 6
  How many shoulder flexions (0-90 degrees), in a given pace, with a 3 kg (men) or 2 kg (women) dumbbell in the hand is possible to do
Self-reported disease activity | Baseline, months 3 and 6
  The patient-reported questionnaire Systemic Lupus Erythematosus Activity Questionnaire includes three parts. The part about disease symptoms goes from 0-47 points, the higher the points the more disease symptoms. Further there is a question about flares with four answer alternatives, from no flares to serious flares. There is also a numerical rating scale about disease activity on a scale from 0-10, the higher value the higher the disease activity
Fatigue | Baseline, months 3 and 6
  The patient-reported questionnaire Functional Assessment of Chronic Illness Therapy, FACIT-Fatigue goes from 0-52 points, the higher the value, the less the fatigue
Anxiety and depressive symptoms | Baseline, months 3 and 6
  The patient-reported questionnaire Hospital Anxiety and Depression scale goes from 0-21 points, the higher the value, the higher the anxiety and depressive symptoms. In the anxiety and depressive symptoms subscales the points goes from 0-6, the higher the value, the higher anxiety and depressive symptoms respectively
Quality of life in SLE | Baseline, months 3 and 6
  The patient-reported questionnaire Lupus Quality of life questionnaire goes from 0-100 points, the higher the value the better the quality of life
Generic Quality of life | Baseline, months 3 and 6
  The patient-reported questionnaire Short Form Health Survey (SF-36). Each subscale goes from 0-100 points, the higher the value, the higher the quality of life.
Quality of life and health status | Baseline, months 3 and 6
  The patient-reported questionnaire EuroQol 5-dimensions (EQ-5D). The index scores goes from -0,594 till 1,000, the higher the value, the higher the quality of life
Disease activity | Baseline, months 3 and 6
  SLE Disease Activity Index 2000 (SLEDAI-2K) assessed by a physician, goes from 0-105 points, the higher the value, the higher the disease activity
Inflammatory markers | Baseline, months 3 and 6
  Blood samples are collected before and after maximal ergometercycle exercise test
Health status | Baseline, months 3 and 6
  The patient-reported questionnaire EuroQol 5-dimensions (EQ-5D)-5L Visual analogue scale, 0-100 mm, the higher the value, the better the health
Blood pressure | Baseline, month 3 and 6
  Resting diastolic and systolic blood pressure

OTHER OUTCOMES:
Organ damage | Baseline and 6 months
  Systemic Lupus International Collaborating Clinics (SLICC/ACR-Damage Index). Organ damage last 6 months, assessed by a physician. The points goes from 0-47, the higher the value, the more organ damage
Demographical, clinical and lifestyle behaviour data including age, gender, ethnic origin, and smoking status as well as other for the project important information about the disease such as autoantibody profiles and pharmacological treatment | Baseline. For some variables, such as medical treatment, also months 3 and 6
  A questionnaire developed specific for this project and data from patients medical files
Physical activity | Baseline, months 3 and 6
  The patient-reported questionnaire International Physical Activity Questionnaire addresses the number of days and time spent on physical activity in moderate intensity, vigorous intensity and walking of at least 10-min duration the last 7 days, and also includes time spent sitting on weekdays the last 7 days. The sum score is expressed in physical activity Metabolic Equivalent of Task-minutes per day or week
Activity-minutes and sitting behaviour | Baseline, months 3 and 6
  The patient-reported questions about Activity-minutes and sitting behaviour according to the Swedish National Board of Health and Welfare. For the two questions about physical training and exercise with 5 respective 6 answer alternatives, the higher the value, the more time spending training and exercising. The question about sitting have 7 answer alternatives, the higher the value, the less time spent sitting
Weight | Baseline, months 3 and 6
  Weight in kilograms
Height | Baseline
  Height in meters
Body Mass Index (BMI) | Baseline, months 3 and 6
  Weight in kilograms divided by the height in metres squared
Muscle function lower extremity | Baseline, months 3 and 6
  How many times is it possible to raise from a chair during 30 seconds; the "30 seconds Chair stand test"

CONTACTS AND LOCATIONS:
Overall Officials: Carina M Boström, Dr, Principal Investigator — Karolinska Institutet
Locations (1):
- Carina Boström, Stockholm, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: No